CLINICAL TRIAL: NCT00622973
Title: Noninvasive Detection of Clinically Occult Lymph Node Metastases in Prostate and Bladder Cancer Evaluated by USPIO-Enhanced MRI and Diffusion-Weighted MRI: A Histopathological Correlation
Brief Title: USPIO-enhanced and Diffusion-weighted MRI for the Detection of Pelvic Lymph Node Metastases
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Harriet C. Thoeny, MD, University Hospital Inselspital, Berne
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: SNF320000-113512/1; KEK101_06; SNF320000-113512/1; SWISSMEDIC2007DR3215
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Prostate Cancer; Bladder Cancer
Keywords: Prostate cancer; Bladder cancer; Pelvic lymph node metastases; Diffusion-weighted MRI; Sinerem (USPIO)-enhanced MRI; Imaging influence on surgery; Noninvasive detection of pelvic lymph node metastases; Influence of imaging protocol on surgical outcome
MeSH Terms: conditions — Prostatic Neoplasms; Urinary Bladder Neoplasms | interventions — ferumoxtran-10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other): Diffusion-weighted MRI
  Interventions: Other: Imaging: diffusion-weighted MRI
- B (Other): Sinerem (USPIO)- enhanced MRI
  Interventions: Other: Sinerem (USPIO) enhanced MRI

INTERVENTIONS:
Other: Imaging: diffusion-weighted MRI — Diffusion-weighted MRI of the entire pelvis to detect lymph node metastases
  Arms: A
Other: Sinerem (USPIO) enhanced MRI — USPIO (Sinerem) will be administered intravenously immediately after the first MR examination at a dose of 2.6 mg Fe/kg body weight diluted in 100 ml of saline (optimal dose according to: (9, 10)) during a period of about 30 minutes under medical supervision. Postcontrast MR imaging will be performed 24-36 hours after contrast medium injection.
  Other Names: SINEREM
  Arms: B

SUMMARY:
Preoperative detection of lymph node metastases in patients with prostate or bladder cancer is crucial for selection of the appropriate treatment strategy (surgery, androgen deprivation with/or without radiation therapy or chemotherapy) and thus for patient prognosis. Until now CT or MRI have been the modalities of choice for preoperative staging procedures. However, current morphological assessment of lymph nodes based on size and shape is unable to detect smaller metastases or liable to give false positive results on lymph nodes with reactive hyperplasia. We hypothesize that USPIO-enhanced MRI combined with DW-MRI will be able to detect pelvic lymph node metastases preoperatively with high sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven prostate cancer (T1-2N0M0 Gleason score 6-10) scheduled for radical prostatectomy or patients with histologically proven bladder cancer (T1-3bN0M0G3) scheduled for cystectomy
* Written informed consent to participate in this trial.

Exclusion Criteria:

* Patients with contraindications for MRI (e.g. pacemaker, metal implants, claustrophobia).
* Patients in a critical cardiovascular state, with risk of decompensation after administration of the USPIO contrast agent.
* Patients with hemochromatosis or an allergy to dextran or iron compounds.
* Pregnant or breast-feeding women.
* Patients who have received gadolinium complexes within 2 days or iron oxide particles within 7 days before MRI.
* Patients who underwent chemotherapy or radiotherapy before surgery.
* Patients whose degree of cooperation is incompatible with carrying out the study.
* Patients with contraindications to Glucagon administration.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2007-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Discrimination of N positive (N+) vs. N negative (N0) patients (prostate and bladder cancer) using diffusion-weighted imaging, USPIO enhancement and both. | 1 year
Preoperative localization of all suspected positive nodes in accordance to the predefined regions on both sides and in comparison with histopathology. | 1 year

SECONDARY OUTCOMES:
Node-by-node analysis of USPIO-enhanced and DW-MRI positive lymph nodes with histopathology. | 2-3 years

CONTACTS AND LOCATIONS:
Overall Officials: Harriet C Thoeny, MD, Principal Investigator — University Hospital Inselspital, Bern, Switzerland
Locations (1):
- Inselspital, Bern, Switzerland

REFERENCES:
- [Result] Thoeny HC, Triantafyllou M, Birkhaeuser FD, Froehlich JM, Tshering DW, Binser T, Fleischmann A, Vermathen P, Studer UE. Combined ultrasmall superparamagnetic particles of iron oxide-enhanced and diffusion-weighted magnetic resonance imaging reliably detect pelvic lymph node metastases in normal-sized nodes of bladder and prostate cancer patients. Eur Urol. 2009 Apr;55(4):761-9. doi: 10.1016/j.eururo.2008.12.034. Epub 2009 Jan 7. PMID 19144456
- [Derived] Birkhauser FD, Studer UE, Froehlich JM, Triantafyllou M, Bains LJ, Petralia G, Vermathen P, Fleischmann A, Thoeny HC. Combined ultrasmall superparamagnetic particles of iron oxide-enhanced and diffusion-weighted magnetic resonance imaging facilitates detection of metastases in normal-sized pelvic lymph nodes of patients with bladder and prostate cancer. Eur Urol. 2013 Dec;64(6):953-60. doi: 10.1016/j.eururo.2013.07.032. Epub 2013 Jul 30. PMID 23916692
- [Derived] Triantafyllou M, Studer UE, Birkhauser FD, Fleischmann A, Bains LJ, Petralia G, Christe A, Froehlich JM, Thoeny HC. Ultrasmall superparamagnetic particles of iron oxide allow for the detection of metastases in normal sized pelvic lymph nodes of patients with bladder and/or prostate cancer. Eur J Cancer. 2013 Feb;49(3):616-24. doi: 10.1016/j.ejca.2012.09.034. Epub 2012 Oct 18. PMID 23084842